CLINICAL TRIAL: NCT05067608
Title: Study on the Safety and Efficacy of Cryopreserved Platelets in Hypoproliferative Thrombocytopenic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: DSO National Laboratories (Other); Health Sciences Authority, Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPPL-DSO-2018; 2018/2883 (Other: Centralised Institutional Review Board (CIRB))
Record Dates: First submitted 2021-08-02; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Hypoproliferative Thrombocytopenia
Keywords: Hypoproliferative thrombocytopenia; Cryopreserved; Transfusion; Platelets; Safety; Efficacy
MeSH Terms: interventions — Platelet Count

STUDY DESIGN:
Intervention Model Description: This is a phase 1b/2a single centre clinical trial. Eligible hypoproliferative thrombocytopenic adult patients enrolled in the study will be randomised into two arms. One arm is the "treatment" arm using cryopreserved platelets and the second is the "control" arm using liquid platelets. A recruitment period of two years is expected for 17 subjects in each arm. Subjects will automatically be crossed over to the other treatment arm once they have completed the first treatment arm and there is at least a 5-days interval without platelet transfusion. Subjects can be both inpatient and outpatient. During the thrombocytopenic period of 28 days, subjects may be required to have multiple platelet transfusions during this period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Subjects in the "control" arm will receive normal pooled platelets for all of their transfusion within a single thrombocytopenic period. If subjects participate in the study for more than one thrombocytopenic period, they will automatically be enrolled in the opposing arm for their second thrombocytopenic period.
  Interventions: Biological: Control arm receiving normal (never before frozen) platelets as per current clinical practice
- Treatment arm (Experimental): Subjects in the "treatment" arm will receive thawed cryopreserved pooled platelets for all of their transfusions (except for unplanned or urgent platelet transfusions outside stipulated periods when thawed cryopreserved platelets are unavailable) within a single thrombocytopenic period. If subjects participate in the study for more than one thrombocytopenic period, they will automatically be enrolled in the opposing arm for their second thrombocytopenic period.
  Interventions: Biological: Treatment arm receiving cryopreserved platelets

INTERVENTIONS:
Biological: Control arm receiving normal (never before frozen) platelets as per current clinical practice — Liquid platelets arm (control) and may receive multiple platelet transfusions per thrombocytopenic cycle.
  Arms: Control arm
Biological: Treatment arm receiving cryopreserved platelets — Cryopreserved platelets arm (treatment) and may receive multiple platelet transfusions per thrombocytopenic cycle.
  Arms: Treatment arm

SUMMARY:
The purpose of this study is to study the safety and efficacy of pooled buffy-coat derived platelets which had been frozen with dimethyl sulphoxide (DMSO), in the prevention of bleeding for patients with hypoproliferaitve thrombocytopenia. These platelets are hereafter referred to as cryopreserved platelets. Patients who have severely low platelet count due to impaired bone marrow function from chemotherapy or certain haematological conditions may need platelet transfusion to prevent spontaneous bleeding. Currently, platelets are stored in liquid form, and must be used within five to seven days of collection. In this study, DMSO is used to preserve platelets during freezing so that they can be stored for longer than five to seven days. Investigators hope to learn if thawed cryopreserved platelets are functional and safe for transfusion in humans.

DETAILED DESCRIPTION:
Platelets are currently stored in liquid form for a maximum of five to seven days. To extend the shelf-life of platelets, DMSO is added to freeze platelets for long-term storage. In vitro studies have shown that such cryopreserved platelets can be kept for at least two years at -80oC. This study is a clinical trial that aims to primarily assess the safety of cryopreserved pooled buffy coat-derived platelets in patients with hypoproliferative thrombocytopenia and no platelet refractoriness.

Subjects will be randomised into two arms either a liquid platelet (control) or frozen platelet arm (treatment) and may receive four or more platelet transfusions per thrombocytopenic cycle. Each subject may participate in the study for up to two thrombocytopenic period, assuming a wash-out period of at least five days (during which the subject receives no platelet transfusions) between the two thrombocytopenic periods. If subjects participate in the study for more than one thrombocytopenic period, they will automatically be enrolled in the opposing arm for their second thrombocytopenic period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 21 years of age
2. Be able to provide written informed consent
3. Current or potential hypoproliferative thrombocytopenia with expected platelet count of <20 X 109/L for a minimum of 5 days in a 28-day period
4. If pre-menopausal female of child bearing potential, then the subject must have a negative serum pregnancy test prior to study commencement, and must be using an acceptable method of contraception during the study.
5. Calculated creatinine clearance of >30 ml/min (as calculated based on the Cockcroft-Gault equation; National Kidney Foundation 2017) at the point of recruitment, and within one week before transfusion

Exclusion Criteria:

1. Not meeting the inclusion criteria specified above
2. Pregnant
3. Breastfeeding
4. Current platelet refractoriness
5. History of allergy or adverse reaction to DMSO
6. History of veno-occlusive disease
7. History of acute venous or arterial thromboembolism within the last 3 months.
8. History of unprovoked venous thromboembolism
9. On antiplatelets, NSAIDs or anticoagulants within 1 week, and TCM (traditional Chinese medicine) which are known to decrease platelet count or platelet function or increase bleeding tendency within 2 weeks of study enrolment.
10. Received or will be receiving L-asparaginase chemotherapy within 7 days of platelet transfusion
11. Renal impairment with calculated creatinine clearance of <30ml/min.
12. Non-cutaneous Grade 2 and above bleeding at the time of study assessment
13. Presently with or a history of acute promyelocytic leukemia (APML), immune thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), haemolytic-uremic syndrome (HUS), or any thrombotic microangiopathy (TMA)
14. Presently with or a history of heparin-induced thrombocytopenia
15. Presently with disseminated intravascular coagulation (DIC) or other risk factor(s) for bleeding other than thrombocytopenia (including platelet dysfunction, PT ≥ 1.3 X upper limit of normal for the laboratory, PTT ≥ 1.3 X upper limit of normal for the laboratory, or fibrinogen ≤ 1 g/L)
16. History of anaphylaxis from blood transfusion
17. Involved in any other therapeutic clinical trials in the last 6 months prior to the start of this research
18. Concomitant participation in other therapeutic clinical trials during the full period of this study
19. Receiving non-trial-related medication that might compromise transfusion safety
20. Known history of congenital bleeding disorder
21. Subject who declined to consent for platelet transfusion

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to platelet transfusion. | Monitoring will be for 24 hours (serum test 18-30 hours) post-transfusion.
  There would be a close visual observation of the patient throughout the transfusion for the earliest signs of a transfusion reaction. Because patients can experience transfusion reactions several hours after the transfusion is completed, inpatients should be observed for late reactions during the subsequent 24 hour. Outpatient patients and their carer would be counselled about the possibility of the late adverse reactions and given access to immediate clinical help if they develop any symptoms of a transfusion reaction within 24 hour post-transfusion. Patients receiving cryopreserved platelets will be monitored and assessed for the side-effects of DMSO within 24 hour. These side effects include: headache, nausea, sedation, dizziness, abdominal or chest & abdominal discomfort during and after transfusion. It also includes assessment for renal impairment related to DMSO by performing serum renal panel 18 to 30 hours post-transfusion of study platelets.
Non-cutaneous Grade 2 or higher bleeding (as defined on the WHO bleeding scale) | Each thrombocytopenic period is up to 28 days from the first prophylactic platelet transfusion (shorter if platelet count recovers above target level before 28 days)
  Patients will be monitored daily for bleeding during each thrombocytopenic period if they are inpatients. If they are outpatients, they will be reviewed for bleeding at each clinic visit, and they will be asked to keep a record of any bleeding symptoms which will also be reviewed at each clinical visit during each of the thrombocytopenic periods.

SECONDARY OUTCOMES:
Platelet count increase (absolute increase and corrected count increment) post-platelet trantrsfusion | Within approximately 24 hours prior, 1-4 hour and 18-30 hour post-transfusion.
  A pre-transfusion (baseline) venous blood sample for FBC will be taken by a trained phlebotomist/ nurse using Vacutainer tubes from the subject approximately within 24 hours prior to the planned platelet transfusion (for both "control" and "treatment" arms). Post-transfusion venous blood sample for FBC will be taken by a trained phlebotomist or nurse using Vacutainer tubes form the subject at 1-4 hour and 18-30 hour after transfusion.
Changes in platelet activity (measured by viscoelastic hemostatic assay) post-platelet transfusion | Within approximately 24 hours prior, 1-4 hour and 18-30 hour post-transfusion.
  A pre-transfusion (baseline) venous blood sample for VHA (viscoelastic hemostatic assay) will be taken by a trained phlebotomist/ nurse using Vacutainer tubes from the subject approximately within 24 hours prior to the planned platelet transfusion (for both "control" and "treatment" arms). Post-transfusion venous blood sample for VHA will be taken by a trained phlebotomist or nurse using Vacutainer tubes form the subject at 1-4 hour and 18-30 hour after transfusion.
Changes in procoagulant activity post-platelet transfusion | Within approximately 24 hours prior and 1-4 hour post-transfusion.
  A pre-transfusion (baseline) venous blood sample for procoagulant assays will be taken by a trained phlebotomist/ nurse using Vacutainer tubes from the subject approximately within 24 hours prior to the planned platelet transfusion (for both "control" and "treatment" arms). Post-transfusion venous blood sample for procoagulant assays will be taken by a trained phlebotomist or nurse using Vacutainer tubes form the subject at 1-4 hour after transfusion.
Incidence of all grades of bleeding (as defined on WHO bleeding scale) | Each thrombocytopenic period is up to 28 days from the first prophylactic platelet transfusion of each arm (shorter if platelet count recovers above target level before 28 days)
  Patients will be monitored daily for bleeding during each thrombocytopenic period if they are inpatients. If they are outpatients, they will be reviewed for bleeding at each clinic visit, and they will be asked to keep a record of any bleeding symptoms which will also be reviewed at each clinical visit during each of the thrombocytopenic periods.
Total number and type of blood products transfused | Each thrombocytopenic period is up to 28 days from the first prophylactic platelet transfusion of each arm (shorter if platelet count recovers above target level before 28 days)
  For each thrombocytopenic period, subject may receive platelets and other types of blood components.
  The time and type of blood components administered (including the non-study ones) would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ang Ai Leen, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Will not be sharing individual participant data collected in this study to other researchers.

REFERENCES:
- [Background] ClinicalTrials.gov: NCT02078284. Phase 1 safety study of dimethyl sulphoxide cryopreserved platelets.
- [Background] Dumont LJ, Dumont DF, Unger ZM, Siegel A, Szczepiorkowski ZM, Corson JS, Jones MK, Christoffel T, Pellham E, Bailey SL, Slichter SJ; BEST Collaborative. A randomized controlled trial comparing autologous radiolabeled in vivo platelet (PLT) recoveries and survivals of 7-day-stored PLT-rich plasma and buffy coat PLTs from the same subjects. Transfusion. 2011 Jun;51(6):1241-8. doi: 10.1111/j.1537-2995.2010.03007.x. Epub 2011 Jan 7. PMID 21214584
- [Background] Dumont LJ, Cancelas JA, Graminske S, Friedman KD, Vassallo RR, Whitley PH, Rugg N, Dumont DF, Herschel L, Siegal AH, Szczepiorkowski ZM, Fender L, Razatos A. In vitro and in vivo quality of leukoreduced apheresis platelets stored in a new platelet additive solution. Transfusion. 2013 May;53(5):972-80. doi: 10.1111/j.1537-2995.2012.03841.x. Epub 2012 Aug 6. PMID 22882530
- [Background] Noorman F, van Dongen TT, Plat MJ, Badloe JF, Hess JR, Hoencamp R. Transfusion: -80 degrees C Frozen Blood Products Are Safe and Effective in Military Casualty Care. PLoS One. 2016 Dec 13;11(12):e0168401. doi: 10.1371/journal.pone.0168401. eCollection 2016. PMID 27959967
- [Background] Slichter SJ, Jones M, Ransom J, Gettinger I, Jones MK, Christoffel T, Pellham E, Bailey SL, Corson J, Bolgiano D. Review of in vivo studies of dimethyl sulfoxide cryopreserved platelets. Transfus Med Rev. 2014 Oct;28(4):212-25. doi: 10.1016/j.tmrv.2014.09.001. Epub 2014 Sep 21. PMID 25439164